CLINICAL TRIAL: NCT01802099
Title: Impact of Early Enteral vs. Parenteral Nutrition on Mortality in Patients Requiring Mechanical Ventilation and Catecholamines: Multicenter, Randomized Controlled Trial (NUTRIREA-2)
Brief Title: Impact of Early Enteral vs. Parenteral Nutrition on Mortality in Patients Requiring Mechanical Ventilation and Catecholamines
Acronym: NUTRIREA2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped on Data Safety and Monitoring Board 's request
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHD085-11
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure; Shock
Keywords: mechanical ventilation; early enteral nutrition; intensive care unit; early parenteral nutrition; critical care medicine; nosocomial infection; mortality; shock; vasoactive drug
MeSH Terms: conditions — Shock; Hyperphagia; Cross Infection | interventions — Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenteral nutrition (Other): Patients will receive parenteral nutrition during the first week of mechanical ventilation. After Day 3, the parenteral route may be switched to the enteral route if shock resolve (vasoactive drug stopped since 24 hours and serum lactate level < 2 mmol/l). After Day 7, all patients will be fed via the enteral route.
  Interventions: Other: Parenteral nutrition
- Enteral nutrition (Other): Patients will receive nutrition only via the enteral route during the firs week of invasive mechanical ventilation.
  Interventions: Other: Enteral nutrition

INTERVENTIONS:
Other: Enteral nutrition
  Other Names: Enteral feeding
  Arms: Enteral nutrition
Other: Parenteral nutrition
  Other Names: Intravenous nutrition; intravenous feeding
  Arms: Parenteral nutrition

SUMMARY:
The purpose of this study is to assess the hypothesis that, as compared to early intravenous feeding, early nutrition via the enteral route is associated with reduced Day 28-mortality in critically ill patients treated with mechanical ventilation and vasoactive drug.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation expected to be required more than 48 hours
* Nutrition started within 24 hours after initiation of endotracheal mechanical ventilation
* Treatment with vasoactive drug administered via a central venous catheter
* Age over 18 years
* Signed information

Exclusion Criteria:

* Abdominal surgery within 1 month before inclusion
* History of esophageal, gastric, duodenal or pancreatic surgery
* Bleeding from the esophagus, stomach or bowel
* enteral nutrition via gastrostomy or jejunostomy
* pregnancy
* Treatment-limitation decisions
* Current inclusion in a trial on comparison between enteral and parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2411 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Reignier, MD, PhD, Principal Investigator — CHD Vendee
Locations (41):
- France (41):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - Centre hospitalier d'Annecy, Annecy
  - Centre Hospitalier de Beauvais, Beauvais
  - CHU Besançon-Hôpital Jean Minjoz, Besançon
  - CHU Pellegrin Tripode, Bordeaux
  - CH Louis Pasteur, Chartres
  - CHU Gabriel Montpied, Clermont Ferrand, Clermont-Ferrand
  - CHU Louis Mourier, Colombes
  - CH de Dieppe, Dieppe
  - CHU Dijon, Dijon
  - Hôpital Raymond Poincarre, Garches
  - CHU Grenoble, Grenoble
  - CHD Vendée - service de réanimation, La Roche-sur-Yon
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - CH Docteur Schaffner, Lens
  - CHU Lille, Lille
  - CHU de Lyon- Hôpital de la Croix Rousse, Lyon
  - Hospices Civils de Lyon, Lyon
  - CH Marc Jacquet, Melun
  - CH de Montauban, Montauban
  - CHI André Grégoire, Montreuil
  - Hôpital Emile Muller, Mulhouse
  - CHU de Nantes, Hopital Laennec, Nantes
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Hôpital de La Source, CHR Orléans, Orléans
  - CHU Saint Louis, Paris
  - CHU Saint-Antoine, Paris
  - CHU Paris Cochin, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - Hôpital Tenon, Paris
  - CHU Pointe à Pitre - Abymes, Pointe à Pitre
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Jacques Puel, Rodez
  - Hôpital Delafontaine, Saint-Denis
  - CHU Saint Etienne-Hôpital Nord, Saint-Etienne
  - CH de Saint Malo, St-Malo
  - CHU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Tours, Tours

REFERENCES:
- [Background] Brisard L, Le Gouge A, Lascarrou JB, Dupont H, Asfar P, Sirodot M, Piton G, Bui HN, Gontier O, Hssain AA, Gaudry S, Rigaud JP, Quenot JP, Maxime V, Schwebel C, Thevenin D, Nseir S, Parmentier E, El Kalioubie A, Jourdain M, Leray V, Rolin N, Bellec F, Das V, Ganster F, Guitton C, Asehnoune K, Bretagnol A, Anguel N, Mira JP, Canet E, Guidet B, Djibre M, Misset B, Robert R, Martino F, Letocart P, Silva D, Darmon M, Botoc V, Herbrecht JE, Meziani F, Devaquet J, Mercier E, Richecoeur J, Martin S, Greau E, Giraudeau B, Reignier J. Impact of early enteral versus parenteral nutrition on mortality in patients requiring mechanical ventilation and catecholamines: study protocol for a randomized controlled trial (NUTRIREA-2). Trials. 2014 Dec 23;15:507. doi: 10.1186/1745-6215-15-507. PMID 25539571
- [Result] Reignier J, Boisrame-Helms J, Brisard L, Lascarrou JB, Ait Hssain A, Anguel N, Argaud L, Asehnoune K, Asfar P, Bellec F, Botoc V, Bretagnol A, Bui HN, Canet E, Da Silva D, Darmon M, Das V, Devaquet J, Djibre M, Ganster F, Garrouste-Orgeas M, Gaudry S, Gontier O, Guerin C, Guidet B, Guitton C, Herbrecht JE, Lacherade JC, Letocart P, Martino F, Maxime V, Mercier E, Mira JP, Nseir S, Piton G, Quenot JP, Richecoeur J, Rigaud JP, Robert R, Rolin N, Schwebel C, Sirodot M, Tinturier F, Thevenin D, Giraudeau B, Le Gouge A; NUTRIREA-2 Trial Investigators; Clinical Research in Intensive Care and Sepsis (CRICS) group. Enteral versus parenteral early nutrition in ventilated adults with shock: a randomised, controlled, multicentre, open-label, parallel-group study (NUTRIREA-2). Lancet. 2018 Jan 13;391(10116):133-143. doi: 10.1016/S0140-6736(17)32146-3. Epub 2017 Nov 8. PMID 29128300

RESULTS

PARTICIPANT FLOW:
Groups:
- Parenteral Nutrition: Patients will receive parenteral nutrition during the first week of mechanical ventilation. After Day 3, the parenteral route may be switched to the enteral route if shock resolve (vasoactive drug stopped since 24 hours and serum lactate level < 2 mmol/l). After Day 7, all patients will be fed via the enteral route.
  Parenteral nutrition
- Enteral Nutrition: Patients will receive nutrition only via the enteral route during the firs week of invasive mechanical ventilation.
  Enteral nutrition
Period: Overall Study
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Started | 1208 | 1202
Completed | 1208 | 1202
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parenteral Nutrition | Enteral Nutrition | Total
Number analyzed (Participants) | 1208 | 1202 | 2410
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (14) | 66 (14) | 66 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 815 | 809 | 1624
  Male | 393 | 393 | 786
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 1208 | 1202 | 2410

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Number analyzed (Participants) | 1208 | 1202
Participants | 422 | 443

2. Secondary Outcome: Mortality Rate
Time Frame: 90 days
Reporting Status: Not Posted

3. Secondary Outcome: Ventilator-associated Pneumonia Rate
Time Frame: until weaning of mechanical ventilation (average: 7 days)
Reporting Status: Not Posted

4. Secondary Outcome: Nosocomial Infections Rate
Description: Bloodstream infection Urinary tract infection Catheter-related infection Other infections
Time Frame: until discharge from ICU (average: 10 days)
Reporting Status: Not Posted

5. Secondary Outcome: Length of Stay in Intensive Care Unit (ICU)
Time Frame: until discharge from ICU (average: 10 days)
Reporting Status: Not Posted

6. Secondary Outcome: Length of Stay in Hospital
Time Frame: until discharge from hospital (average: 17 days)
Reporting Status: Not Posted

7. Secondary Outcome: Variations in Sepsis-related Organ Failure Assessment (SOFA) Score
Time Frame: first week (7 days) of mechanical ventilation
Reporting Status: Not Posted

8. Secondary Outcome: Calories Intake
Time Frame: until weaning of mechanical ventilation (average : 7 days)
Reporting Status: Not Posted

9. Secondary Outcome: Proportion of Patients Given 100% of the Calorie Target
Time Frame: until weaning of mechanical ventilation (average: 7 days)
Reporting Status: Not Posted

10. Secondary Outcome: Cumulative Calorie Deficit From Day 0 to Day 7
Time Frame: During the first week (7 days) of mechanical ventilation
Reporting Status: Not Posted

11. Secondary Outcome: Hospital Mortality Rate
Time Frame: Until discharge from hospital (average : 17 days)
Reporting Status: Not Posted

12. Secondary Outcome: Intensive Care Unit (ICU) Mortality Rate
Time Frame: until discharge from ICU (average: 10 days)
Reporting Status: Not Posted

13. Secondary Outcome: Acute Bowel Ischemia Rate
Time Frame: until weaning of mechanical ventilation (average: 7 days)
Reporting Status: Not Posted

14. Secondary Outcome: Vomiting Rate
Time Frame: until weaning of mechanical ventilation (average: 7 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Parenteral Nutrition | Enteral Nutrition
Serious Adverse Events (participants affected / at risk) | 0/1208 | 0/1202
Other Adverse Events (participants affected / at risk) | 0/1208 | 0/1202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT01802099/Prot_SAP_000.pdf